CLINICAL TRIAL: NCT03792464
Title: Serum Hepcidin and Iron Status Parameters in Pregnant Women and the Association With Adverse Maternal and Fetal Outcome
Brief Title: Serum Hepcidin in Pregnant Women and the Association With Pregnancy Outcome
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-02322
Record Dates: First submitted 2018-12-03; First posted 2019-01-03 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Hematological and serum iron parameters will be determined using routine laboratory methodology. Blood samples are collected by venipuncture. All blood measurements will be conducted at the University Hospital of Basel, Department of Laboratory Medicine.
  Hb, RBC, HCT, MCV, MCHC, MRC, HRC and CHr are measured using a hematology analyzer. Mean corpuscular hemoglobin is automatically calculated from Hb and RBC. Ferritin is assessed by chemiluminescence immunoassay and CRP is assessed by immunoturbidimetry. Soluble transferrin receptors and serum hepcidin are measured with an ELISA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepcidin production is normally upregulated by iron stores, and in obesity has been shown to be overexpressed and correlated with low iron status. The increased hepcidin may restrain the iron release from the cells by affecting the expression of ferroportin, which probably associates with the development of diabetes complication. Firstly, investigator examines the difference of serum hepcidin and iron parameters between obese and non-obese pregnant women; secondly, the correlation between serum hepcidin and adverse maternal and neonatal outcomes in pregnant women will be tested.

DETAILED DESCRIPTION:
This is a mono-center, observational, controlled study with 2 parallel groups (obese versus non-obese pregnant women). The study will be conducted at the University Hospital of Basel, Department of Obstetrics and Antenatal Care. A total of N=188 healthy pregnant women (expected 40% with BMI ≥ 30 kg/m2) will be recruited in the first trimester in our outpatients' department in order to have a total of 169 evaluable women, considering a drop-out rate of 10%. Serum hepcidin, iron and hematological parameters will be measured at 11-14, 24-28, 32-36 weeks of gestation and at labor. The blood pressure, weight, weight gain, BMI and smoking status will be examined at all visits. Blood samples will be measured in the University Hospital of Basel, Department of Laboratory Medicine. Recruitment will begin in January 2019.

ELIGIBILITY:
Inclusion Criteria:

* women with a BMI ≥ 18.5 kg/m2,
* maternal age ≥ 18 years,
* singleton pregnancy,
* gestational age at recruitment: 11-14 of gestational weeks,
* written informed consent.

Exclusion Criteria:

* pregnant women with a BMI< 18.5 kg/m2,
* congenital anomaly of fetus,
* severe maternal diseases of heart, liver, kidney, cardiovascular system, gastrointestinal tract, neurologic disorders and psychiatric disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: 188 singleton pregnancies will be recruited in the first trimester at the University Hospital of Basel, Department of Obstetrics and Antenatal Care.
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Serum hepcidin at 11-14 weeks of gestation | 11-14 weeks of gestation
  serum hepcidin (ng/ml)

SECONDARY OUTCOMES:
Serum hepcidin at 24-28, 32-36 weeks of gestation and at labor; | at 24-28, 32-36 weeks of gestation
  serum hepcidin (ng/ml)
serum ferritin (µg/l), | at 24-28, 32-36 weeks of gestation
  iron status Parameter
HRC (%), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
hemoglobin (g/l), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
red blood cells (x1012/l), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
hematocrit (l/l), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
MCV (fl), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
MCH (pg), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
MCHC (g/l), | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
red blood cell distribution width (%) | at 11-14, 24-28, 32-36 weeks of gestation
  blood parameter
soluble transferrin receptors (mg/l) | at 24-28, 32-36 weeks of gestation
  iron status Parameter

OTHER OUTCOMES:
preeclampsia (presence: yes/no) | from 11 week of gestation to the 3 days after the birth
  maternal outcome
pregnancy induced hypertension (presence: yes/no), | from 11 week of gestation to the birth
  maternal outcome
infection in pregnancy (presence: yes/no), | from 11 week of gestation to the 5 days after the birth
  maternal outcome
anemia (presence: yes/no) | from 11 week of gestation to 3 days after the birth
  maternal outcome
iron deficiency (presence: yes/no), | from 11 week of gestation to the birth
  maternal outcome
cholestasis in pregnancy (presence:yes/no), | from 11 week of gestation to the birth
  maternal outcome
gestational diabetes mellitus (presence: yes/no), | from 11 week of gestation to the birth
  maternal outcome
abnormal placentation (presence: yes/no), | from 11 week of gestation to the birth
  maternal outcome
blood loss during birth (ml) | at the birth
  maternal outcome
transfusion requirement (presence: yes/no) | at the birth
  maternal outcome
gestational age at birth (gestational week and day) | at the birth
  neonatal outcome
birth weight (g) | at the birth
  neonatal outcome
preterm delivery (presence: yes/no) | at the birth
  neonatal outcome
preterm premature rupture of fetal membrane (presence: yes/no) | at the birth
  neonatal outcome
intrauterine growth restriction (yes/no) | from 11 week of gestation to the birth
  neonatal outcome
intrauterine fetal death | from 11 week of gestation to the birth
  neonatal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Amstad Bencaiova, Principal Investigator — Department of Obsterics, University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Amstad G, Geiger J, Werlen L, Montavon C, Heinzelmann V. Perioperative management with ferric carboxymaltose and tranexamic acid to reduce transfusion rate in gynaecological carcinoma surgery (TRANAFER-Study): study protocol for a single-blind, monocentre, randomised trial. BMJ Open. 2022 Sep 26;12(9):e057381. doi: 10.1136/bmjopen-2021-057381. PMID 36167367
- [Derived] Amstad Bencaiova G, Vogt DR, Hoesli I. Serum hepcidin and iron status parameters in pregnant women and the association with adverse maternal and fetal outcomes: a study protocol for a prospective cohort study. BMJ Open. 2019 Nov 6;9(11):e032280. doi: 10.1136/bmjopen-2019-032280. PMID 31699745